CLINICAL TRIAL: NCT02815592
Title: A Phase 1/2 Randomized Trial of BMS-986012 in Combination With Platinum and Etoposide as First-line Therapy in Extensive-Stage Small Cell Lung Cancer
Brief Title: Trial of BMS-986012 in Combination With Platinum and Etoposide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA001-044; 2016-001692-67 (EudraCT Number)
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Cisplatin; Etoposide; Platinum; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Experimental Arm 1 (Experimental): BMS-986012/Cisplatin/Etoposide
  Interventions: Drug: BMS-986012; Drug: Cisplatin; Drug: Etoposide
- Experimental Arm 2 (Experimental): BMS-986012/Carboplatin/Etoposide
  Interventions: Drug: BMS-986012; Drug: Etoposide; Drug: Carboplatin
- Experimental Arm 3A (Experimental): BMS-986012/Platinum/Etoposide
  Interventions: Drug: BMS-986012; Drug: Etoposide; Drug: Platinum
- Active Comparator Arm 3B (Active Comparator): Platinum/Etoposide
  Interventions: Drug: Etoposide; Drug: Platinum

INTERVENTIONS:
Drug: BMS-986012
  Arms: Experimental Arm 1; Experimental Arm 2; Experimental Arm 3A
Drug: Cisplatin
  Arms: Experimental Arm 1
Drug: Etoposide
Drug: Platinum
  Arms: Active Comparator Arm 3B; Experimental Arm 3A
Drug: Carboplatin
  Arms: Experimental Arm 2

SUMMARY:
The purpose of this this study is to administer BMS-986012 in Combination with Platinum and Etoposide as First-line Therapy in Extensive Small Cell Lung Cancer.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Male and Females 18 years of age or older
* Pulmonary SCLC documented by histology or cytology
* Extensive disease (Stage IV) SCLC
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

* Prior systemic therapy for lung cancer
* Symptomatic brain metastases
* Grade 2 peripheral neuropathy
* Active or chronic infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV
* Other active malignancies or prior malignancy within 2 years

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Cycle 1, Day 1 up to approximately 26 months.
Number of participants with serious adverse events (SAEs ) | Date of enrollment up to approximately 26 months.
Discontinuations due to AEs | Cycle 1, Day 1 up to approximately 26 months.
Number of participants who died due to AEs | Cycle 1, Day 1 up to approximately 26 months.
Number of participants with laboratory toxicity grade shift from baseline | Cycle 1, Day 1 up to approximately 26 months.
Progression Free Survival | From date of first dose or randomization until date of confirmed disease progression, up to 2 years

SECONDARY OUTCOMES:
Maximum observed serum concentration(Cmax) | Cycle 1 Day 1 up to 60 days after last dose
Time of maximum observed serum concentration(Tmax) | Cycle 1 Day 1 up to 60 days after last dose
Area under the plasma concentration-time curve from time 0 to time of last quantifiable concentration(AUC(0-T)) | Cycle 1 Day 1 up to 60 days after last dose
Observed serum concentration at the end of a dosing interval(Ctau) | Cycle 1 Day 1 up to 60 days after last dose
Area under the concentration-time curve in 1 dosing interval(AUC(TAU)) | Cycle 1 Day 1 up to 60 days after last dose
Characterization of Immunogenicity | Cycle 1 Day 1 up to 60 days after last dose
  Anti-Drug Antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- Spain (4):
  - Local Institution - 0002, Barcelona
  - Local Institution - 0004, Madrid
  - Local Institution - 0003, Majadahonda - Madrid
  - Local Institution - 0010, Málaga

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/home